CLINICAL TRIAL: NCT05801107
Title: A Phase II Study to Investigate the Efficacy and Safety of WX-0593 in Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: Study to Investigate the Efficacy and Safety of WX-0593 in ALK Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-007
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX0593 (Experimental): 60 mg of WX-0593 tablets, once daily for 7 days, followed by 180 mg of WX-0593 tablets, once daily in a 21-days cycle.
  Interventions: Drug: WX-0593

INTERVENTIONS:
Drug: WX-0593 — WX-0593 Tablets 60 mg QD，once daily for 7 days, followed by 180 mg of WX-0593 tablets,once daily in a 21-days cycle.
  Other Names: FL-006

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of WX-0593 in patients with ALK-positive NSCLC

ELIGIBILITY:
Key Inclusion Criteria:

* ≥18 years
* Female or male
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of at least 12 weeks
* At least one measurable lesion
* Histologically or cytologically confirmed diagnosis of advanced or recurrent or metastatic NSCLC that is ALK-positive by grade A tertiary hospitals, and subjects should have disease progression (RECIST 1.1) or intolerance (stopping criteria according to drug insert) after 1 or 2 marketed ALK inhibitors, the patients had disease progression after ALK inhibitor should continuously have drug at least 12 weeks , and less than 3 chemotherapy regimens previously
* No brain metastasis, or asymptomatic brain metastasis, or symptomatic brain metastasis but stable for more than 4 weeks after treatment, and have stopped systemic hormone treatment (prednisone of > 10 mg/day or equivalent hormone) for more than 2 weeks

Key Exclusion Criteria:

* Crizotinib is the only ALK inhibitor subjects received;unmarketed ALK inhibitor received; Lorlatinib or Brigatinib received; active ingredient or generic drug of ALK inhibitors received
* HBsAg-positive and/or HBcAb positive and HBV DNA > 1000 copies/mL, or HCV antibody-positive, or known HIV infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Assessed By independent radiology review | From first administration to the date that the last patients observed for 18 weeks
  ORR is defined the percentage of the participants who have achieved complete response (CR) or partial response (PR) per independent radiology review using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, PhD, Study Chair — Shanghai Jiao Tong University Chest Hospital
Locations (1):
- Shanghai Jiao Tong University Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No